CLINICAL TRIAL: NCT01562847
Title: Dynamics of ABL Mutations in Imatinib Failed Ph Positive or Bcr-Abl Positive CML CP or AP Patients Who Treated With Nilotinib as Second-line TKI Therapy (AMICAN-Prospective)in Asia
Brief Title: Prospective Investigation of Dynamics of ABL Mutations in Imatinib Failed CML Patients Treated With Nilotinib
Acronym: AMICAN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Dong-Wook Kim, Professor, Seoul St. Mary's Hospital
Other Study IDs: CAMN107AKR05T
Record Dates: First submitted 2011-07-21; First posted 2012-03-26 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA analysis for mutation and Bcr-Abl gene quantification using mainly peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nilotinib
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Patients will be treated with 800 mg nilotinib daily.
  Other Names: Nilotinib: Tasigna

SUMMARY:
The purposes of this study are to investigate expression and frequency of ABL point mutations, a major cause of resistance in imatinib failed CML Asian patients and to find causes of Asian-specific resistance to cancer-targeting therapies through a prospective investigation of dynamics of point mutations and expression of new point mutations during nilotinib treatment.

DETAILED DESCRIPTION:
Recently the treatment strategy of Philadelphia chromosome-positive leukemia has undergone groundbreaking changes due to the development of new second-generation cancer-targeting drugs. After 2001, a seven-year survival for leukemia stands at as much as 86 percent due to the oral therapy of cancer-targeting imatinib as a standard treatment, but drug resistance occurs in some patients in the early stage of the treatment. It is known that weakened binding ability of imatinib to BCR-ABL is due to a point mutation in the ATP-binding site of BCR-ABL. This accounts for 70 percent of causes of imatinib resistance. According to the studies so far, there are approximately more than 60 types of BCR-ABL point mutation, which causes imatinib resistance.

The international phase II clinical study of dasatinib and nilotinib, second-generation cancer-targeting therapies, in imatinib failed patients which began in 2005 showed that more than 70 percent of the patients achieved a complete hematological response (CHR) again, and about 50 percent of the patients, a major hematological response (MHR). In the study, it was also observed that kinase activation was inhibited by a second-generation cancer-targeting therapy for most of the major imatinib-resistant point mutations. With regard to peculiar point mutations, V299L, F317L, and E25K/V show relative resistance to dasatinib, and p-loop mutations including G250E, Q252H, Y253F/H and E255K/V and F359C/V show relative resistance to nilotinib. T315I mutation exhibits strong resistance to both of these cancer-targeting therapies. Therefore, it is considered that the second-generation cancer-targeting therapies show therapeutic effects in different domains.

According to the results of the recent studies including the one conducted by our center, it is assumed that imatinib resistance caused by point mutations in patients induces more point mutations and causes selective increase in T315I point mutations during treatment of the second-generation cancer-targeting therapy.

However, in the studies so far, the subjects were selectively chosen in advance for the pharmaceutical company to receive an approval from the health authorities and ABL point mutations were followed up during the limited study period, which indicates that there have been limits to accurately observe and evaluate dynamics of point mutations throughout treatment with the second-generation cancer-targeting drug.

For this reason, this study is designed to examine ABL point mutations in patients with Philadelphia chromosome-positive or BCR-ABL-positive chronic leukemia who are treated with imatinib, to observe dynamics of existing point mutations during treatment with nilotinib, and to confirm the mechanism of resistance including expression of new point mutations and their expression patterns through a long-term follow-up. In addition, this study will confirm whether expression pattern of ABL point mutations associated with nilotinib in Asian is different from that in Western patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia chromosome-positive or BCR-ABL positive CML
* Chronic, Accelerated phase CML patients who show an inappropriate response to the imatinib treatment or failed the treatment according to ELN 2009 RECOMMENDATION
* Patients with ECOG performance status of 0-3
* Patients who consent to the use of study information and study specimen

Exclusion Criteria:

* Patients with diseases other than CML
* Patients treated with myelosuppressive anticancer therapy other than Hydroxyurea and Angrelide
* Patients who have been treated with second-generation cancer-targeting drug
* Patients who do not consent to the use of study information and study specimen
* Previously documented T315I mutation
* Impaired cardiac function including any of the following: LVEF by echocardiography < 45% or below the institutional lower range (whichever is greater); complete left bundle branch block; long QT syndrome or family history of; history or presence of significant ventricular or atrial tachyarrhythmias; clinically significant brachycardia (< 50 bpm); QTcF > 450 msec at baseline; right bundle branch block plus left anterior hemiblock; bifascicular block; myocardial infarction ≤ 12 months; uncontrolled angina; other clinically significant heart disease (e.g., congestive heart failure)
* Treatment with strong inhibitors of CYP3A4 or medication that are well documented to prolong the QT interval are contraindicated
* Impaired gastrointestinal(GI)function or GI disease that may significantly alter the absorption of the study drug (e.g., ulcerative diseases, uncontrolled nausea, vomitting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery)
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* Know cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required)
* Patients who previously had a bone marrow or stem cell transplantation
* Pregnant or breast-feeding patients
* Hypersensitivity to nilotinib or any of the excipients
* The capsules contain lactose, and nilotinib is therefore not recommended for patients with rare hereditary problem of galactose intolerance, severe lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean Adult CML patients
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
To confirm the patterns of resistance including point mutations which are newly expressed during the nilotinib treatment | 5 years

SECONDARY OUTCOMES:
To analyze and evaluate the overall survival and disease free survival in the nilotinib treatment according to progression of the disease and types of point mutations | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wook Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea